CLINICAL TRIAL: NCT03885362
Title: Assessment of the Accuracy of Continuous Glucose Sensors in People With Diabetes Undergoing Haemodialysis
Acronym: ALPHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18SM4938
Record Dates: First submitted 2019-02-22; First posted 2019-03-21 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Diabetic Nephropathies; Type 1 Diabetes Mellitus; Chronic Kidney Diseases
Keywords: Type 1 Diabetes Mellitus; Chronic Kidney Diseases
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 1; Renal Insufficiency, Chronic

STUDY DESIGN:
Masking Description: Blinded CGM but not Libre
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dexcom G6 and Abbott Freestyle Libre (Experimental): Participants will have a Dexcom G6 sensor and Abbott FreeStyle Libre sensor inserted in the abdomen and upper arm respectively. Participants will be asked to swipe the FreeStyle Libre reader across the sensor a minimum of every 8 hours. Participants will be asked to continue their usual regimen of self-monitoring capillary blood glucose (SMBG).
  During haemodialysis, a dialysis circuit blood sample will be drawn at 0 (pre-dialysis) 30, 60, 90, 120, 150, 180, 210 and 240 minutes and immediately after dialysis. Samples from the circuit will be analysed on the YSI glucose analyser. Participants will be asked to change the FreeStyle Libre sensors at day 14. The blinded CGM data will be uploaded at the time of each sensor change by the research team.
  Interventions: Device: Dexcom G6 and Abbott Freestyle Libre

INTERVENTIONS:
Device: Dexcom G6 and Abbott Freestyle Libre — Dexcom G6 - continuous glucose monitoring device - blinded. CE mark 2018 Abbott Freestyle Libre - flash glucose monitoring device. CE mark 2014

SUMMARY:
The purpose of the study is to assess the accuracy of the Dexcom G6 CGM system and the Abbott FreeStyle Libre flash system compared to the reference standard YSI (Yellow Spring Instruments) glucose in people with diabetes undergoing haemodialysis. The Dexcom G6 is a continuous glucose monitoring system that gives blood glucose values in real-time and includes alarms if the glucose is very low or high. The Abbott FreeStyle ibre flash system is an intermittent glucose monitor that shows the blood glucose values when it is waved near the sensor and does not include alarms. The YSI glucose analysis will take place as a normal part of haemodialysis, by testing blood glucose levels during the haemodialysis session. The study will last 28 days per participant

DETAILED DESCRIPTION:
Diabetic nephropathy is the leading cause of end-stage renal failure (ESRF), representing approximately 40% of people requiring long-term renal replacement therapy and maintenance haemodialysis [1]. Mortality and morbidity within this cohort is high, with the predominant cause being cardiovascular disease (CVD) [2]. Glycaemic control in many haemodialysis dependent patients with diabetes is poor and may lead to additional renal complications, including high interdialytic weight gain, electrolyte imbalance, and amputations [3]. Current clinical guidance is centred around the prevention of hyperglycaemia and microvascular complications of diabetes.

Glucose self-management is particularly challenging due to cyclical changes in insulin sensitivity and circulating insulin concentrations. Hypoglycemia is common due to impaired renal gluconeogenesis, malnutrition, and the increased half-life of insulin and hypoglycemic agents [4, 5]. Additionally, people with chronic kidney disease and diabetes may have other diabetes complications such as retinopathy, neuropathy, and impaired awareness of hypoglycaemia, which can make self-management more difficult.

Overall assessment of glycaemic control is also more complex as classical markers of glycemic control (i.e. HbA1c and fructosamine) may be misleading due to the variable underestimation of glycaemia resulting from analytical interferences, shortened half-life of red blood cells and abnormal albumin level [6-8]. Further limitations of HbA1c is that it is not informative regarding glycemic control on the days on and off dialysis, and intra-day glycaemic variability.

Frequent capillary blood glucose tests or self-monitoring of blood glucose (SMBG) is the traditional and one of the most effective ways to track an individuals' blood glucose levels. Real-time continuous glucose monitoring (CGM) has been shown to improve overall glucose control, reduce hypoglycaemia in people with an HbA1c <7.0%, and may reduce severe hypoglycaemia [9-11]. In addition, they provide alert and alarm features for hypo- and hyperglycaemia, and for times of rapid glucose change.

Flash glucose monitoring does not provide real-time data with alerts and alarms, but allows users to retrospectively review the preceding 8 hours of continuous glucose data, along with a contemporary estimated blood glucose value and trend line. The system consists of a subcutaneous sensor placed on the back of the upper arm, which measures glucose in the interstitial fluid every minute. The glucose data are made available when the user chooses to swipe the reader over the sensor.

CGM has the potential to reduce HbA1c and minimize exposure to hypoglycaemia while addressing diabetes distress. Flash glucose monitoring may reduce exposure to hypoglycaemia in people with insulin-treated diabetes.

The accuracy of CGM and flash in people with diabetes on haemodialysis has not been described. In this clinical study, the investigators will assess the accuracy of the Dexcom G6 CGM system and the Abbott FreeStyle Libre flash system compared to YSI (Yellow Spring Instruments) glucose in people undergoing haemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years of age
* Diabetes, with insulin treatment for over 6 months or on sulphonylureas
* Chronic kidney disease requiring haemodialysis three times per week

Exclusion Criteria:

* Pregnant or planning pregnancy
* Breastfeeding
* Enrolled in other clinical trials
* Have active malignancy or under investigation for malignancy
* Severe visual impairment
* Reduced manual dexterity
* Unable to participate due to other factors, as assessed by the Chief Investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-11 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
MARD between G6 and YSI | 28 days
  Mean absolute relative difference between Dexcom G6 and YSI glucose during haemodialysis
MARD between Libre and YSI | 28 days
  Mean absolute relative difference between Dexcom G6 and YSI glucose during haemodialysis

SECONDARY OUTCOMES:
HbA1c | 28 days
  Glycated Haemoglobin
MARD for G6 and YSI <3.9mmol/L | 28 days
  Mean absolute relative difference between Dexcom G6 and YSI glucose <3.9mmol/L
MARD for Libre and YSI <3.9mmol/L | 28 days
  Mean absolute relative difference between Libre and YSI glucose <3.9mmol/L
MARD for Libre and YSI 3.9-10mmol/L | 28 days
  Mean absolute relative difference between Libre and YSI glucose 3.9-10mmol/L
MARD for Libre and YSI >10mmol/L | 28 days
  Mean absolute relative difference between Libre and YSI glucose >10mmol/L
MARD for G6 and YSI 3.9-10mmol/L | 28 days
  Mean absolute relative difference between Dexcom G6 and YSI glucose 3.9-10mmol/L
MARD for G6 and YSI >10mmol/L | 28 days
  Mean absolute relative difference between Dexcom G6 and YSI glucose >10mmol/L
MARD for G6 and YSI 24hr pre | 24 hours
  Mean absolute relative difference between Dexcom G6 and YSI glucose during 24 hours prior to heamodialysis
MARD for Libre and YSI 24hr pre | 24 hours
  Mean absolute relative difference between Libre and YSI glucose during 24 hours prior to heamodialysis
MARD for Libre and YSI 24hr post | 24 hours
  Mean absolute relative difference between Libre and YSI glucose during 24 hours after heamodialysis
MARD for G6 and YSI 24hr post | 24 hours
  Mean absolute relative difference between Dexcom G6 and YSI glucose during 24 hours after heamodialysis
CEG analysis G6 and YSI | 28 DAYS
  Clarke Error Grid analysis between Dexcom G6 and YSI glucose during haemodialysis
CEG analysis Libre and YSI | 28 DAYS
  Clarke Error Grid analysis between Libre and YSI glucose during haemodialysis
Severe hypoglycaemia | 28 days
  Episodes of severe hypoglycaemia
DKA | 28 days
  Diabetic Ketoacidosis
Sensor failure | 28 days
  Events of G6/libre sensor failure
Missing glucose data | 28 days
  Missing blood glucose data for G6/libre measured by number of missing data points

CONTACTS AND LOCATIONS:
Overall Officials: Nick Oliver, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London/NHS trust Renal Unit, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coresh J, Selvin E, Stevens LA, Manzi J, Kusek JW, Eggers P, Van Lente F, Levey AS. Prevalence of chronic kidney disease in the United States. JAMA. 2007 Nov 7;298(17):2038-47. doi: 10.1001/jama.298.17.2038. PMID 17986697
- [Background] Levin A. Clinical epidemiology of cardiovascular disease in chronic kidney disease prior to dialysis. Semin Dial. 2003 Mar-Apr;16(2):101-5. doi: 10.1046/j.1525-139x.2003.16025.x. PMID 12641872
- [Background] Creme D, McCafferty K. Glycaemic Control Impact on Renal Endpoints in Diabetic Patients on Haemodialysis. Int J Nephrol. 2015;2015:523521. doi: 10.1155/2015/523521. Epub 2015 Sep 20. PMID 26457201
- [Background] National Kidney Foundation. KDOQI Clinical Practice Guideline for Diabetes and CKD: 2012 Update. Am J Kidney Dis. 2012 Nov;60(5):850-86. doi: 10.1053/j.ajkd.2012.07.005. PMID 23067652
- [Background] Haviv YS, Sharkia M, Safadi R. Hypoglycemia in patients with renal failure. Ren Fail. 2000 Mar;22(2):219-23. doi: 10.1081/jdi-100100866. PMID 10803766
- [Background] Lee KF, Szeto YT, Benzie IF. Glycohaemoglobin measurement: methodological differences in relation to interference by urea. Acta Diabetol. 2002 Apr;39(1):35-9. doi: 10.1007/s005920200010. PMID 12043937
- [Background] Inaba M, Okuno S, Kumeda Y, Yamada S, Imanishi Y, Tabata T, Okamura M, Okada S, Yamakawa T, Ishimura E, Nishizawa Y; Osaka CKD Expert Research Group. Glycated albumin is a better glycemic indicator than glycated hemoglobin values in hemodialysis patients with diabetes: effect of anemia and erythropoietin injection. J Am Soc Nephrol. 2007 Mar;18(3):896-903. doi: 10.1681/ASN.2006070772. Epub 2007 Jan 31. PMID 17267743
- [Background] Joy MS, Cefalu WT, Hogan SL, Nachman PH. Long-term glycemic control measurements in diabetic patients receiving hemodialysis. Am J Kidney Dis. 2002 Feb;39(2):297-307. doi: 10.1053/ajkd.2002.30549. PMID 11840370
- [Background] Pickup JC, Freeman SC, Sutton AJ. Glycaemic control in type 1 diabetes during real time continuous glucose monitoring compared with self monitoring of blood glucose: meta-analysis of randomised controlled trials using individual patient data. BMJ. 2011 Jul 7;343:d3805. doi: 10.1136/bmj.d3805. PMID 21737469
- [Background] Beck RW, Riddlesworth T, Ruedy K, Ahmann A, Bergenstal R, Haller S, Kollman C, Kruger D, McGill JB, Polonsky W, Toschi E, Wolpert H, Price D; DIAMOND Study Group. Effect of Continuous Glucose Monitoring on Glycemic Control in Adults With Type 1 Diabetes Using Insulin Injections: The DIAMOND Randomized Clinical Trial. JAMA. 2017 Jan 24;317(4):371-378. doi: 10.1001/jama.2016.19975. PMID 28118453
- [Background] Lind M, Polonsky W, Hirsch IB, Heise T, Bolinder J, Dahlqvist S, Schwarz E, Olafsdottir AF, Frid A, Wedel H, Ahlen E, Nystrom T, Hellman J. Continuous Glucose Monitoring vs Conventional Therapy for Glycemic Control in Adults With Type 1 Diabetes Treated With Multiple Daily Insulin Injections: The GOLD Randomized Clinical Trial. JAMA. 2017 Jan 24;317(4):379-387. doi: 10.1001/jama.2016.19976. PMID 28118454